CLINICAL TRIAL: NCT04418401
Title: A Study on the Safety and Efficacy of Donafinib Combined With Anti-PD-1 Antibody as Adjuvant Therapy for HCC Patients With High Risks of Recurrence
Brief Title: Study on the Safety and Efficacy of Donafinib Combined With Anti-PD-1 Antibody as Adjuvant Therapy for HCC Patients
Acronym: CISLD-8
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Proffessor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CISLD-8
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Postoperation; High risk of recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Treatment with Donafenib 100mg PO BID，and anti-PD-1 antibody 3mg/kg ivgtt Q2W. Treatment will last 6 months, unless the tumor recurrence.
  Interventions: Drug: Donafenib and anti-PD-1 antibody

INTERVENTIONS:
Drug: Donafenib and anti-PD-1 antibody — Donafenib was taken orally twice daily, and anti-PD-1 antibody was applied biweekly.

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignant tumors, with more than 700,000 new cases in the world every year. China has the highest incidence and death rate of HCC in the world, accounting for 55% of the world's annual incidence and 45% of the world's annual deaths. At present, surgical resection is still one of the most effective treatments for HCC. However, the recurrence rate of tumor after hepatectomy is still very high, and the recurrence rate of 5 years is 60~70%. Especially in patients with high-risk recurrence factors, without intervention, the cumulative recurrence rate in the first year was about 50%, about 60% in the second year, about 70% in the third year, and about 80% in the fifth year. Tumor recurrence is an important bottleneck that hinders the long-term survival of patients. Therefore, there is an urgent need for effective adjuvant therapy to reduce the postoperative recurrence rate of patients with HCC, especially high-risk patients. However, there is still a lack of standard protocols for postoperative adjuvant therapy for HCC. Here investigators intend to explore the safety and efficacy of Donafinib Combined With Anti-PD-1 Antibody as postoperative adjuvant therapy for HCC patients with high risks of recurrence.

DETAILED DESCRIPTION:
This is a single center, open, single arm, and exploratory study. Thirty HCC patients with high risk recurrence factors after radical surgery will be enrolled. Adjuvant treatment of Donafenib combined with anti-PD-1 antibody will be given for 6 months. The primary endpoint is the cumulative percentage of patients without recurrence in the first year. The recurrence-free survival (RFS), overall survival (OS), tumor recurrence time (TTR), ECOG physical condition (ECOG PS) score, the changes of FACT-Hep based quality of life score, changes of AFP, and adverse events will be recorded and analyzed, to evaluated the efficacy and safety of this combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1)Voluntary admission and signature of written informed consent;

2)18~75 years of age (including 75 years), male and female;

3)Hepatocellular carcinoma underwent radical resection 4~8 weeks before enrolled.

4)Pathologically diagnosed as hepatocellular carcinoma with any of the following conditions: a)Microvascular invasion (MVI); b)Satellite nodules were found in specimens; c)Multiple tumor nodules(>3 nodules); d)Portal vein tumor thrombosis (PVTT): The tumor thrombosis invades the left or right branches of portal vein, with or without hepatic vein invasion;

5)≥4 weeks after radical resection, the imaging examination confirmed no recurrence and metastasis.

6)Liver function Child-Pugh grade A (5~6);

7)Physical condition was scored 0~1 according to the ECOG criteria.

8)Expected lifetime >3 months;

9)HBV DNA<10^4 copy/ ml (2000 IU/ ml); if HBV DNA ≥10^4 copy/ ml, antiviral therapy should be given, until the HBV DNA drops below 10^4Copy/ml patient can be enrolled in the study. And during the study, antiviral drugs should be continued, and liver function and hepatitis B virus load should be monitored;

10)The results of the serum pregnancy test must be negative for women with fertility (i.e. non-menopausal or surgical sterilization) within 7 days prior to the study of drug administration;

11)The main organs function normally: Blood routine examination (no transfusion, no use of G-CSF within 14 days before screening): a)Hemoglobin ≥90 g/L; b)Absolute neutrophil count (ANC)≥1.5×10^9/L; c)Platelet count ≥75×10^9/L; Blood biochemical examination (albumin not used within 14 days before screening): d)Albumin ≥28 g/L; e)Total bilirubin ≤1.5× ULN; f)Aspartate aminotransferase (AST), alanine aminotransferase (ALT )≤3× ULN; g)Serum creatinine ≤1.5×ULN; Coagulation function: h)The international standardized ratio (INR) or prothrombin time (PT )≤1.5×ULN;. i)Activated partial thromboplastin time (APTT )≤1.5×ULN.

Exclusion Criteria:

1. Histopathological diagnosis of hepatocellular carcinoma - intrahepatic cholangiocarcinoma (HCC-ICC) mixed type;
2. Positive resection margin or tumor rupture;
3. Operation of recurrent liver cancer;
4. Other malignancies within 5 years unless the patient has received a possible cure and there is no evidence of the disease within 5 years, but this time requirement (i.e. within 5 years) is not applicable to patients with skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ or other carcinoma in situ who have successfully undergone excision;
5. Previous or present congenital or acquired immunodeficiency disease;
6. Active or previously documented autoimmune or inflammatory diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, pituitary inflammation, hyperthyroidism or hypothyroidism, asthma requiring treatment with bronchiectasis, etc.), asthma with vitiligo or which has been completely relieved in childhood without inclusion of any intervention in adults;
7. History of severe mental illness;
8. Suffer from diseases (e.g. severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorders, etc.) that affect the absorption, distribution, metabolism or clearance of the study drug;

   Past or combined medication/treatment:
9. Had major surgery (defined by the investigators) within 4 weeks before admission, or expected to require major surgery during study therapy;
10. Previous transplantation of allogeneic stem cells or parenchymal organs;
11. Preoperative treatment with sorafenib, valvatinib, regofenib or immunomodulator such as anti PD-1、 PD-L1、 anti CTLA-4;
12. Patients who have received other systemic anti-tumor treatments before surgery, including traditional Chinese medicine with anti-tumor indications, have had less than 2 weeks or 5 half-time (whichever is longer) between the completion of the treatment and the use of the drugs before the study, or who have not recovered to ≤CTCAE 1 level of adverse events caused by preoperative treatment;
13. Other adjuvant therapy (except antiviral therapy) was performed after operation.
14. Systemic immunosuppressive drugs have been used within 2 weeks before admission or are expected to be required during the study period, except in the following cases: a)Intra-nasal, inhalation, topical or topical (e.g. intra-articular) corticosteroids; b)Prednisone ≤ 10 mg/day or other equivalent systemic corticosteroid; c)Prophylactic use of corticosteroids for hypersensitivity;
15. Take drugs that may prolong QTc and/or induce advanced torsional ventricular tachycardia (Tdp) or affect drug metabolism;
16. Patients with known or suspected history of allergies to Donafenib or similar drugs, hypersensitivity to chimeric or humanized antibodies or fusion proteins, or to excipients used to study drugs;
17. The presence of uncontrollable hepatic encephalopathy, hepatorenal syndrome, ascites, pleural effusion or pericardial effusion;
18. Active bleeding or abnormal coagulation function, bleeding tendency or undergoing thrombolytic, anticoagulant or antiplatelet therapy;
19. There was a history of gastrointestinal bleeding or a definite tendency of gastrointestinal bleeding in the past 4 weeks (e.g. local active ulcer lesions, stool occult blood≥ ++ , e.g. continuous stool occult blood +, gastroscopy should be performed), or other conditions (e.g. severe gastric fundus/esophageal varices) that the researchers determined might cause gastrointestinal bleeding;
20. Gastrointestinal perforation, abdominal fistula or abdominal abscess occurred within 6 months.
21. Thrombosis or thromboembolic events, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc., occurred within 6 months.
22. With significant clinical significance, including but not limited to previous 6 months of acute myocardial infarction, severe/unstable angina, or coronary artery bypass grafting, congestive heart failure (New York Heart Association NYHA Grade > Grade 2), Poor control or arrhythmia requiring pacemaker therapy, Uncontrolled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg);
23. Active infections, including: a)HIV (HIV 1/2 antibody) positive; b)Active hepatitis B (HBsAg positive and abnormal liver function); c)Active hepatitis C (HCV antibody positive or HCV RNA≥10^3 copy/ ml and abnormal liver function); d)Active tuberculosis; e)Other uncontrolled active infections (CTCAE V5.0> level 2);
24. Other significant clinical and laboratory abnormalities, the researchers believe affect safety evaluation, such as: uncontrolled diabetes, chronic kidney disease, peripheral neuropathy (CTCAE V5.0) of grade II or above, thyroid dysfunction, etc.
25. Has not recovered from surgery, such as the presence of unhealed incisions or severe postoperative complications;
26. Received any live attenuated vaccine within 4 weeks of admission or during the study period;
27. Pregnant or lactating women, as well as women or men with fertility who are unwilling or unable to take effective contraception;
28. A history of alcohol, psychotropic or other substance abuse within 6 months;
29. Enrolled in other clinical trials within 4 weeks before admission.
30. Failure to follow the study protocol for treatment or scheduled follow-up;
31. Any other factors evaluated by investigators that patients cannot be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free rate in one year | Through the study period, for 3 years
  The cumulative percentage of patients without recurrence in the first year after the primary surgery

SECONDARY OUTCOMES:
Recurrence-free survival | Through the study period, for 3 years
  The period from the first study treatment to disease recurrence
Overall survival | Through the study period, for 3 years
  The period from the first study treatment to any cause of death
ECOG physical condition 8/5000 ECOG physical condition | Through the study period, for 3 years
  The changes of physical condition evaluated according to the criteria of Eastern Cooperative Oncology Group
FACT-Hep QLQ | Through the study period, for 3 years
  The change of the quality of life
Alpha fetoprotein | Through the study period, for 3 years
  The change of AFP
Adverse effects | Through the study period, for 3 years
  Adverse events occurring through the study treatment, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No